CLINICAL TRIAL: NCT01968018
Title: A Study of Safety and Efficacy of Ultracet in Patients With Chronic Cancer Pain
Brief Title: A Study of Safety and Effectiveness of Ultracet in Patients With Chronic Cancer Pain
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Janssen-Cilag Ltd.,Thailand (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR013510; TRAMAPANA4001 (Other: Janssen-Cilag Ltd.,Thailand)
Record Dates: First submitted 2013-10-18; First posted 2013-10-23 (Estimated); Last update posted 2013-10-23 (Estimated); Status verified 2013-10

CONDITIONS: Cancer
Keywords: Cancer; Chronic Cancer Pain; Tramadol HCI; Acetaminophen; Analgesics; Pain assessment
MeSH Terms: conditions — Neoplasms | interventions — Ultracet

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Tramadol HCI + acetaminophen (Experimental)
  Interventions: Drug: Tramadol HCI/acetaminophen

INTERVENTIONS:
Drug: Tramadol HCI/acetaminophen — Participants will receive tablet of tramadol HCI (37.5 mg)/acetaminophen (325 mg) on Day 1. Participants may increase their daily dosage of study medication is 1 to 2 tablets every 4 to 6 hours as needed for pain relief up to maximum of 8 tablets per day.
  Other Names: Ultracet

SUMMARY:
The purpose of this study is to evaluate the analgesic (painkiller) effectiveness and safety of combination of tramadol HCI (37.5 mg)/acetaminophen (325 mg) in the treatment of chronic cancer pain.

DETAILED DESCRIPTION:
This is an open-label (all people know the identity of the intervention) study. A total of 35 participants will be enrolled in this study. Participants will receive tablet of combination of tramadol HCI (37.5 mg)/acetaminophen (325 mg) on Day 1. Participants may increase their daily dosage of study medication as 1 to 2 tablets every 4 to 6 hours as needed for pain relief, up to maximum of 8 tablets per day. Rescue medication consisting of Extra Strength Tylenol (500 mg) 2 tablets daily for the first six days of the Open-label Phase will be allowed so that the total daily dose of acetaminophen will not exceed 4,000 mg. The total duration of the study treatment for each participant will be approximately 6 weeks. Safety will be evaluated by assessment of adverse events, clinical laboratory tests, skin site assessments, vital signs, and physical examination which will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Participants whose pain has reached a stage now requiring treatment with a weak opioid, according to the opinion of treating physician
* Participants who have received a regular weak opioid, for at least 48 hours and at a dosage appropriate for their pain at that time
* Participants with a histologically, radiologically or hematologically confirmed malignancy; whose pain is judged by the investigator to be caused by the malignancy

Exclusion Criteria:

* Participants who have already received regular treatment with a strong opioid for their cancer pain. This should not exceed more than 3 doses of a strong immediate release opiod in last 7 days, and none in last 24 hours
* Participants with significant abnormalities in hepatic or renal function which would in the opinion of the investigator, prevent the participants involvement in the study
* Participants with a history of allergy or hypersensitivity to tramadol or acetaminophen
* Participants who, at entry have treatments planned which may alter abruptly, the degree or nature of pain experienced (eg radiotherapy, neurological techniques surgery)
* Participants with a history of abuse of opioid analgesics prior to their diagnosis of cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2004-07; Primary Completion 2007-04 (Actual); Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
Change From Baseline in Brief Pain Inventory (BPI) Pain Severity "Pain at Its Worst" (BPI Item 3) at Day 42 | Baseline (Day 1) to Day 42
  Change from baseline in pain severity was assessed using the Brief Pain Inventory (BPI) questionnaire, specifically "pain at its worst" (BPI item 3) at week 4. Scores could have ranged from 0 to 10, where 0 = no pain and 10 = pain as bad as you can imagine. Negative change from baseline scores indicate improvement in "pain at its worst".
Change from Baseline in Analgesic Effect as Assessed by Brief Pain Inventory (BPI) Item 5 Score | Baseline (Day 1) to Day 42
  The analgesic effect was assessed by the Brief Pain Inventory (BPI) item 5 "pain on average" using a 0 to 10 numeric rating scale, with 0 being "no pain" and 10 being "pain as bad as you can imagine". Higher scores indicate worsening.
Number of Participants With Adverse Events | Up to Day 42
  An adverse event is any untoward medical event that occurs in a participant administered an investigational product, and it does not necessarily indicate only events with clear causal relationship with the relevant investigational product.
Number of Doses of Rescue Medication Over Time | Days 7, 14, 28, 35 and 42
  Number of doses of rescue medication over time were assessed. Rescue medications are medicines that are administered to the participants when the efficacy of the study medication is not satisfactory, or the effect of the study medication is too great and is likely to cause a hazard to the participant, or to manage an emergency situation. Supplemental analgesics (medication used to control pain) were used as rescue medication.

SECONDARY OUTCOMES:
Number of Participants With Patient Global Assessment (PGA) | Day 42
  Participants completed a global assessment with respect to pain control using a 9-point scale (-4 to 4; where, -4=100 percent worse, 0=unchanged and 4=100 percent improvement), safety using 5-point scale (1 to 5; where, 1=no, 2=Mild, 3=Moderate, 4=Severe and 5=most severe side effects) and 5-point overall satisfaction scale (1-5; where, 1=no, 2=mild, 3=moderate, 4=good, 5=excellent).
Number of Participants With Investigator Global Assessment | Day 42
  Investigator completed a global assessment of the participants treatment with respect to pain control using a 9-point scale (-4 to 4; where, -4=100 percent worse, 0=unchanged and 4=100 percent improvement), safety using 5-point scale (1 to 5; where, 1=no, 2=mild, 3=moderate, 4=severe and 5=most severe side effects) and 5-point overall satisfaction scale (1-5; where, 1=no, 2=mild, 3=moderate, 4=good, 5=excellent).
Change From Baseline in Quality of Life (QOL) by Using Functional Assessment of Cancer Therapy General Scale (FACT-G) Total Score at Day 42 | Baseline (Day 1) and Day 42
  FACT-G is the 27 items compilation of general Functional Assessment of Cancer Therapy General Scale questions divided into 4 primary dimension of Quality of life (QOL): Physical Well-Being (PWB; 7 items), Social/Family Well-Being (SFWB; 7 items), Emotional Well-Being (EWB; 6 items) and Functional Well-Being (FWB; 7 items). FACT-G uses 5-point Linkert-type response categories ranging from 0="not at all" to 4="very much" to score. Total FACT-G score is the summation of 4 subscale scores and ranges from 0-108. Higher scores for the scales and subscales indicate better QOL.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen-Cilag Ltd.,Thailand Clinical Trial, Study Director — Janssen-Cilag Ltd.,Thailand
Locations (1):
- Bangkok, Thailand